CLINICAL TRIAL: NCT03716024
Title: A Randomized, Evaluator-Blinded, Phase 2 Study to Compare the Safety and Efficacy of PTK 0796 With Linezolid (Zyvox®) in the Treatment of Adults With Complicated Skin and Skin Structure Infection (cSSSI)
Brief Title: Study the Efficacy and Safety of PTK 0796 in Patients With Complicated Skin and Skin Structure Infection (CSSSI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTK0796-CSSI-0702
Record Dates: First submitted 2018-10-17; First posted 2018-10-23 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Infectious Skin Disease; Bacterial Skin Disease
Keywords: CSSSI
MeSH Terms: conditions — Skin Diseases, Infectious; Skin Diseases, Bacterial | interventions — 7-dimethylamino-9-(2,2-dimethylpropyl)aminomethylcycline; Linezolid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PTK 0796 (Experimental)
  Interventions: Drug: PTK 0796
- Linezolid (Active Comparator)
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: PTK 0796 — PTK 0796 100 mg for injection; PTK 0796 capsule 100 mg
  Arms: PTK 0796
Drug: Linezolid — Pre-mixed 600 mg IV infusion solution; Linezolid 600 mg tablets
  Arms: Linezolid

SUMMARY:
A Phase II trial to demonstrate the safety and efficacy of PTK 0796 in the treatment of complicated skin and skin structure infections (cSSSI).

DETAILED DESCRIPTION:
The pharmacologic profile of PTK 0796 in humans suggests that it has the potential to be used safely and effectively for this indication. Data from in vitro and animal studies support this hypothesis.

In PTK 0796-CSSI-0702 the safety and efficacy of PTK 0796 in the treatment of cSSSI will be compared to an antibiotic approved for this indication by FDA. Initial treatment will be administered intravenously with the option for subsequent oral treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, ages 18 years to 80 years
2. Has an acute complicated skin and skin structure infection
3. Female patients must not be pregnant at the time of enrollment and must agree to a reliable method of birth control during the study and for 30 days following the last dose of study drug

Exclusion Criteria:

1. Has received an investigational drug within past 1 month
2. Has been previously enrolled in this protocol
3. Has received >48 hr of a potentially effective systemic antibiotic immediately prior to study drug
4. Is nursing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2007-07-18 (Actual); Primary Completion 2008-01-07 (Actual); Study Completion 2008-01-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Paratek Recruiting Site, Anaheim, California
  - Paratek Recruiting Site, Buena Park, California
  - Paratek Recruiting Site, Chula Vista, California
  - Paratek Recruiting Site, Hawaiian Gardens, California
  - Paratek Recruiting Site, Oceanside, California
  - Paratek Recruiting Site, San Jose, California
  - Paratek Recruiting Site, Indianapolis, Indiana
  - Paratek Recruiting Site, Butte, Montana
  - Paratek Recruiting Site, Electra, Texas
  - Paratek Recruiting Site, Houston, Texas
  - Paratek Recruiting Site, Wichita Falls, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Omadacycline: Participants received intravenous (IV) omadacycline 100 milligrams (mg) infused over 30 minutes, every 24 hours (q24h), with the option to switch to two 100-mg capsules via oral administration q24h at the discretion of the investigator. All participants received up to 7 days of IV therapy and up to 14 days of IV and oral therapy combined.
- Linezolid: Participants received IV linezolid 600 mg infused over 30 minutes, every 12 hours (q12h), with the option to switch to one 600-mg tablet via oral administration q12h at the discretion of the investigator. All participants received up to 7 days of IV therapy and up to 14 days of IV and oral therapy combined.
Period: Overall Study
Arm/Group | Omadacycline | Linezolid
Started | 118 | 116
Completed | 107 | 98
Not Completed | 11 | 18
Not completed — Randomized, not Treated | 7 | 8
Not completed — Adverse Event | 1 | 2
Not completed — Treatment Failure | 1 | 0
Not completed — Lost to Follow-up | 2 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Missing Reason | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for members of the Intent-to-Treat (ITT) Population, comprised of all enrolled participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omadacycline | Linezolid | Total
Number analyzed (Participants) | 111 | 108 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (14.06) | 45.4 (13.34) | 44.9 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 51 | 96
  Male | 66 | 57 | 123
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 97 | 99 | 196
  Black or African American | 8 | 6 | 14
  Asian Hawaiian or Other Pacific Islander | 5 | 1 | 6
  American Indian or Alaska Native | 0 | 1 | 1
  Recorded as Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response in the Modified Intent-to-Treat (mITT) Population
Description: Clinical response is defined as clinical success (CS), which is categorized as a determination by a blinded evaluator (BE) that the infection had sufficiently resolved such that antibiotics were no longer needed, the participant (par.) received ≥1 dose of test article, the par. did not receive non-study antibiotics on >2 calendar days from Day 1 to the Test of Cure assessment, and the par. did not meet any of the criteria for clinical failure. Clinical failure (CF) is categorized as a determination by a BE that the infection had responded inadequately such that alternative antibiotics were needed, the BE discontinued test article due to an adverse event that was possibly/probably related to test article, the primary site of infection was surgically removed, or the par. received potentially effective antibiotics for treatment of the primary infection site on >2 days after study enrollment. A classification of indeterminate is used for any outcome that was not classified as CS or CF.
Time Frame: 10 to 17 days after the last dose of test article (intravenous or oral) (total treatment of up to 14 days)
Population: mITT Population: all enrolled participants who received at least 1 dose of test article and who had at least 1 infecting pathogen isolated at the Baseline evaluation. Non-evaluable participants are included as clinical failures.
Measure: Number; unit: participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 84 | 78
participants
  Clinical success | 75 | 59
  Clinical failure | 9 | 19
  Clinical failure: failure | 2 | 4
  Clinical failure: non-evaluable | 7 | 15
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Superiority; Mean Difference (Final Values) = 13.6, 95% CI 2-sided [1.3 to 26.0] — omadacycline minus linezolid

2. Primary Outcome: Number of Participants With Clinical Response in the Clinically Evaluable (CE) Population
Description: Clinical response is defined as CS, which was categorized as a determination by a BE that the infection had sufficiently resolved such that antibiotics were no longer needed, the participant received ≥1 dose of test article, the participant did not receive non-study antibiotics on >2 calendar days from Day 1 to the Test of Cure assessment, and the participant did not meet any of the criteria for clinical failure. CF was categorized as a determination by a BE that the infection had responded inadequately such that alternative antibiotics were needed, the BE discontinued test article due to an adverse event that was possibly/probably related to test article, the primary site of infection was surgically removed, or the participant received potentially effective antibiotics for treatment of the primary infection site on >2 days after study enrollment. A classification of indeterminate is used for any outcome that was not classified as CS or CF.
Time Frame: 10 to 17 days after the last dose of test article (intravenous or oral) (total treatment of up to 14 days)
Population: CE Population: all enrolled participants who received at least 1 dose of test article and who had a qualifying skin and skin structure infection, received the correct test article for at least 5 calendar days, had the necessary clinical evaluations performed, and did not receive potentially confounding non-study antibiotics
Measure: Number; unit: participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 100 | 88
participants
  Clinical success | 98 | 82
  Clinical failure | 2 | 6
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Superiority; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [-1.7 to 11.4] — omadacycline minus linezolid

3. Secondary Outcome: Number of Participants With Microbiologic Response in the mITT Population
Description: Microbiological response to treatment was determined using the following classification: (a) microbiologic success: all infecting pathogens isolated at Baseline were eradicated or presumed eradicated at the Test of Cure evaluation and no superinfecting pathogen was isolated from the site of infection under study; (b) microbiological failure: persistence or presumed persistence of one or more infecting pathogens or isolation of a superinfecting pathogen from the site of infection under study.
Time Frame: 10 to 17 days after the last dose of test article (intravenous or oral) (total treatment of up to 14 days)
Population: mITT Population. Non-evaluable participants are included as microbiological failures.
Measure: Number; unit: participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 84 | 78
participants
  Microbiological success | 73 | 57
  Microbiological failure | 11 | 21
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Superiority; Mean Difference (Final Values) = 13.8, 95% CI 2-sided [0.9 to 26.7] — omadacycline minus linezolid

4. Secondary Outcome: Number of Participants With Microbiologic Response in the Microbiologically Evaluable (ME) Population
Description: as for outcome 3
Time Frame: 10 to 17 days after the last dose of test article (intravenous or oral) (total treatment of up to 14 days)
Population: ME Population: all participants in the CE cohort who had an infecting pathogen identified at Baseline
Measure: Number; unit: participants
Arm/Group | Omadacycline | Linezolid
Number analyzed (Participants) | 77 | 63
participants
  Microbiological success | 73 | 57
  Microbiological failure | 4 | 6
Statistical Analysis 1: Comparison: Omadacycline vs Linezolid; Test type: Superiority; Mean Difference (Final Values) = 4.3, 95% CI 2-sided [-5.3 to 14.0]

ADVERSE EVENTS:
Time Frame: from enrollment to 10 to 17 days after the last dose of test article (intravenous or oral administration) (up to approximately 27 days)
Description: Adverse events are reported for members of the omadacycline Safety Population, comprised of all participants who received 1 or more doses of omadacycline, and members of the linezolid Safety Population, comprised of all participants who received only linezolid as intravenous test article.
Arm/Group | Omadacycline | Linezolid
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/108
Serious Adverse Events (participants affected / at risk) | 1/111 | 2/108
Other Adverse Events (participants affected / at risk) | 44/111 | 54/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline (N=111) | Linezolid (N=108)
Confusional state (Psychiatric disorders) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline (N=111) | Linezolid (N=108)
Tachycardia (Cardiac disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 13 | 8
Constipation (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 6
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Fatigue (General disorders) | 5 | 2
Abscess (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 0 | 3
Alanine aminotransferase (ALT) increased (Investigations) | 3 | 7
Aspartate aminotransaminase (AST) increased (Investigations) | 3 | 5
Blood creatine phosphokinase increased (Investigations) | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Headache (Nervous system disorders) | 6 | 8
Dizziness (Nervous system disorders) | 4 | 5
Insomnia (Psychiatric disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less